CLINICAL TRIAL: NCT00285545
Title: Biomagnetic Signals of Intestinal Ischemia II
Brief Title: Biomagnetic Signals of Intestinal Ischemia
Status: Completed | Type: Observational
Sponsor: University of South Alabama (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Richards, principal investigator, University of South Alabama
Other Study IDs: DK58197; R01DK058197 (NIH)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Ischemia
Keywords: Blood Supply; Mesentery
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Good blood flow: Group with normal blood flow to small intestine
- Poor blood flow: Group with partial ischemia to small intestine

SUMMARY:
The lack of blood flow to the small intestine causes mesenteric ischemia. Using a Superconducting QUantum Interference Device (SQUID) which measures the magnetic field of the small intestine, we are hoping to identify abnormalities without surgical intervention.

DETAILED DESCRIPTION:
The electrical activity of the small intestine may contain important information that will help us diagnose gastrointestinal diseases. The major impediment to reducing mortality of mesenteric ischemia is the lack of a noninvasive diagnostic test that identifies the syndrome before extensive necrosis occurs. Mesenteric ischemia is caused by the lack of blood flow to the intestine. The Superconducting QUantum Interference Device (SQUID) measures the magnetic field of the intestinal smooth muscle. By comparing normal smooth muscle and that of patients with mesenteric ischemia, we hope to identify abnormal disease states without surgery.

ELIGIBILITY:
Inclusion Criteria:

* Normal Subjects and those diagnosed with mesenteric ischemia

Exclusion Criteria:

* Subjects who report a tendency toward claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2000-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To observe a difference in the magnetic activity between normal and diseased smooth muscle | 2011

CONTACTS AND LOCATIONS:
Overall Officials: William O Richards, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States